CLINICAL TRIAL: NCT00626613
Title: Phase IV Study of General Clinical Research Center Of the Jinan Mental Hospital(TAIWAN)
Brief Title: The Relationship Between Risperdal Treatment and Quality of Life in Patients With Alzheimer's Disease and Behavioural and Psychological Symptoms of Dementia (BPSD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinan Mental Hospital (Other Government)
Collaborators: Johnson & Johnson (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: REM-TWN-MA5
Record Dates: First submitted 2008-02-19; First posted 2008-02-29 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Dementia; Alzheimer's Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Risperidone; Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Risperdal,reminyl — Risperdal:The dosage of treatment medication will begin with 0.5 ml/ per day (0.5mg), The maximum dose will be 2ml/ per day reminyl:8 mg/ per day

SUMMARY:
To evaluate the relationship between Risperidone Treatment, Treatment Discontinuation Rate, and Quality of Life of patients with Alzheimer's Disease and BPSD.

DETAILED DESCRIPTION:
This is an interventional, placebo-controlled, double blind, prospective study. The total duration of this study will be 12 weeks. (1). Baseline Phase: Subjects diagnosed as Alzheimer's Disease and BPSD will be evaluated for entry to the trial. Subjects must meet the inclusion/exclusion criteria before entering the treatment phase. After obtaining informed consent, a physical examination, brief neurologic examination, and clinical laboratory tests appropriate are recommended. (2). Treatment Phase: All patients enrolled will be randomized to treatment with Risperdal Oral Solution or Placebo. The dosage of treatment medication will begin with 0.5 ml/ per day (0.5mg) (as the local product information leaflet). Investigators can titrate dosage according to patients' clinical situation. The maximum dose will be 2ml/ per day. The standardized assessments include NPI, which covers 12 domains of behavioral and neuro-vegetative symptoms, CASI for cognitive function test, and SF-36 for Quality of Life. Adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients whose age 60 years or older diagnosed with Alzheimer's disease and BPSD without exposure to any antipsychotics within 1 month prior to study start.
2. Subjects and subjects' relatives or legal representatives have signed the informed consent form, in accordance with the regulations of the local ethical committee.
3. Subjects must remain in good health, as determined by medical history, complete physical examinations, laboratory tests and ECG.

Exclusion Criteria:

1. Neurodegenerative disorders such as Parkinson's disease, Pick's disease or Huntington's chorea, Down's syndrome, Creutzfeldt-Jacob disease.
2. One of the following conditions possibly resulting in cognitive impairment:

   Acute cerebral trauma caused by post traumatic brain injury, subdural hematoma and injuries secondary to chronic trauma; hypoxic cerebral damage;; cerebral neoplasia;; mental retardation or oligophrenia
3. Multi-infarct dementia or clinically active cerebrovascular disease
4. Subjects with the severe co-existing medical conditions.
5. Current clinically significant cardiovascular disease that would be expected to limit the subject's ability to participate in and complete a 3-month trial.
6. History of drug or alcohol abuse within the last year.
7. Female subjects of childbearing potential without adequate contraception.
8. History of severe drug allergy or hypersensitivity; including recorded hypersensitivity to Risperidone.
9. Participation in a clinical trial of any investigational drug within 1 month (30 days) prior to study entry.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Neoropsychiatric Inventory (NPI)Cognitive Abilities Screening Instrument (CASI) SF-36abnormal involuntary movement scale (AIMS), Barnes akathisia rating scale (BARS), and Simpson angus scale (SAS) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ouyang Wen-Chen, Doctor of Public Health, Principal Investigator — Taiwanese Society of Psychiatry,Boarding member;Zeelandia Dementia Boarding member;Boarding member, Taiwanese Association of Geriatric Psychiatry ;Taiwan Dementia Society Boarding member
Locations (1):
- Department of Psychiatry Jinan Mental Hospital, Tainan, Taiwan